CLINICAL TRIAL: NCT05835401
Title: Effects of Dietary Nitrate Intake on Cardiovascular Performance in Response to Hand Grip Test in Bodybuilders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Cicero Jonas R Benjamim, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: BodyBeet
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Steroid Abuse; Cardiovascular Abnormalities
MeSH Terms: conditions — Cardiovascular Abnormalities | interventions — Nitrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Beetroot juice NO3) (Experimental): Acute ingestion of beetroot juice rich in NO3 (800mg).
  Interventions: Dietary Supplement: Beetroot juice rich in nitrate
- Placebo (Beetroot juice without NO3) (Placebo Comparator): Acute ingestion of beetroot juice rich depleted in NO3.
  Interventions: Dietary Supplement: Beetroot juice depleted in nitrate

INTERVENTIONS:
Dietary Supplement: Beetroot juice rich in nitrate — The participant will intake beetroot juice rich in NO3 (800mg). Two hours after intake the last bottle of juice, the participants will go to the laboratory for the handgrip and cardiovascular tests evaluation. Before crossover protocol a 7-day washout interval will be given for the purification of the compounds provided by the protocols.
  Arms: Experimental (Beetroot juice NO3)
Dietary Supplement: Beetroot juice depleted in nitrate — The participant will intake beetroot juice depleted in NO3. Two hours after intake the last bottle of juice, the participants will go to the laboratory for the handgrip and cardiovascular tests evaluation. Before crossover protocol a 7-day washout interval will be given for the purification of the compounds provided by the protocols.
  Arms: Placebo (Beetroot juice without NO3)

SUMMARY:
Through a randomized, crossover, double-blind, placebo-controlled clinical trial, 20 bodybuilders will participate a acute-day trial with two intervention protocols: 1) placebo and 2) nitrate; in which will ingest beet juice with or without NO3 in its composition with a 7-day washout interval.

ELIGIBILITY:
Inclusion Criteria:

* Anabolic steroid use in the past or actually;
* Participation at least one bodybuilding competition;

Exclusion Criteria:

* Previous history of acute myocardial infarction and/or stroke;
* Allergy or intolerance to nitrate, gluten, or milk;
* Medications (proton pump inhibitors, beta-blockers, calcium channels antagonists).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
1. Values of systolic and diastolic blood pressure (mmHg) | up to 2 years

SECONDARY OUTCOMES:
Plasmatic concentrations of nitrate and nitrite (mmol/L) | up to 2 years
Values of heart rate variability (ms) | up to 2 years
Macrovascular function (Flow mediated dilatation%) | up to 2 years
Values of heart rate (beats per minute) | up to 2 years
Values of hand grip strength (kgF) | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cicero Jonas Rodrigues Benjamim, PhD Student, Principal Investigator — University of Sao Paulo
Locations (1):
- EEFERP - USP / Laboratório de Fisiologia do Exercício e Metabolismo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No